CLINICAL TRIAL: NCT05482828
Title: Effect of Jaeumgeonbi-Tang on Chronic Subjective Dizziness: A Randomized, Double-Blind, Parallel-group, Placebo-Controlled Trial
Brief Title: Effect of Jaeumgeonbi-Tang on Chronic Subjective Dizziness
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The Sponser doesn't fund any more
Sponsor: Korea Health Industry Development Institute (Other Government)
Responsible Party: Principal Investigator, HoRyong Yoo, Associate Professor, Daejeon University, Korea Health Industry Development Institute
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: B100013
Record Dates: First submitted 2013-04-22; First posted 2022-08-01 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Chronic Subjective Dizziness
Keywords: Chronic subjective dizziness; Oxidative stress
MeSH Terms: interventions — Tablets; Starch

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- JGT group (Experimental): Treatment group: JGT (Jaeumgeonbi-Tang) tablet. 8 g t.i.d. for 28 days
  Interventions: Drug: JGT (Jaeumgeonbi-Tang) tablet
- Placebo group (Placebo Comparator): Placebo group: Corn starch tablet, 8 g t.i.d. for 28 days
  Interventions: Drug: Placebo tablet

INTERVENTIONS:
Drug: JGT (Jaeumgeonbi-Tang) tablet — JGT tablet (composed of 19 herbs), 24 g daily (single dose=8 g), t.i.d. for 28 days
  Other Names: JGT (Jaeumgeonbi-Tang) tablet, Hanpoong Co. Ltd
  Arms: JGT group
Drug: Placebo tablet — Corn starch tablet, 24 g daily (single dose=8 g), t.i.d. for 28 days
  Other Names: Corn starch tablet
  Arms: Placebo group

SUMMARY:
The goal of this study is to assess the safety and efficacy of JGT (Jaeumgeonbi-Tang). A randomized, double-blind, parallel-group, placebo-controlled clinical trial was conducted and changes in symptoms and quality of life of the patients were evaluated.

DETAILED DESCRIPTION:
This study's protocol was designed to assess the efficacy of JGT (Jaeumgeonbi-Tang) for chronic subjective dizziness.

* This design of the study is a randomized, double-blind, parallel-group, placebo-controlled design.
* Symptoms and quality of life of chronic subjective dizziness patients will be evaluated.
* Dizziness severity and quality of life of the patients will be evaluated using DHI (Dizziness Handicap Inventory) (1) before treatment (baseline), (2) after 2 weeks, and (3) after 4 weeks of JGT treatment.
* Blood samples of the patients will be gathered before and after JGT treatment for pathophysiological analysis.

ELIGIBILITY:
[Inclusion Criteria]

* Chronic subjective dizziness patients, aged from 20 to 65
* DHI (Dizziness Handicap Inventory) score ≥ 24
* Those who can fully comprehend the general protocol of this study and voluntarily agree to participate

[Exclusion Criteria]

* Inner ear disease (benign paroxysmal positional vertigo, vestibular neuritis, Meniere's disease, etc.)
* Dizziness secondary to specific diseases such as hypoglycemia, recent stroke (within the last 6 months), or heart disease.
* Use of medications that could influence the result of the study (anticonvulsants, sedatives, antidepressants, sleeping pills, prostate medicine, Parkinson's drug, dementia drug, etc.)
* Pregnancy, breastfeeding, or plans of becoming pregnant
* Functional dyspepsia (persistent, recurring abdominal pain, or discomfort)
* Other allergic diseases
* Ineligibility for other reasons in the opinion of the research clinician (when the physician determines that there are significant physical or mental defects that the patient cannot understand and follow the protocol)

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2010-05; Primary Completion 2011-12 (Actual); Study Completion 2013-12-31 (Actual)

PRIMARY OUTCOMES:
Dizziness handicap Inventory | Change from Baseline DHI score at 4 weeks
  The DHI (Dizziness Handicap Inventory) is a 25-item self-report questionnaire that quantifies the effect of dizziness on daily life by measuring the self-perceived handicap of the patients.

CONTACTS AND LOCATIONS:
Overall Officials: Yoo HoRyong, KMD, PhD, Study Director — Daejeon University
Locations (1):
- Daejeon Korean Medicine Hospital of Daejeon Unversity, Daejeon, South Korea

IPD SHARING:
Plan to Share IPD: No